CLINICAL TRIAL: NCT01186796
Title: Role of Endogenous Estrogen in Growth-Hormone Regulation in Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Johannes D. Veldhuis, Johannes D. Veldhuis, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 07-003036
Record Dates: First submitted 2010-08-16; First posted 2010-08-23 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
Keywords: Women; Fulvestrant Study; Post Menopausal Women; Hormones; Healthy Adult Women
MeSH Terms: interventions — Fulvestrant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fulvestrant (Experimental)
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — Secretagogue combinations are assigned in randomized double-blind order within-subject to include the following four conditions:
  (i)L-arginine (30 gm i.v. over 30 min from 0930 h to 1000 h) followed by 5 mL bolus of NS at 1000 h; (ii) L-arginine (30 gm i.v. over 30 min from 0930 h to 1000 h) followed by GHRH and Ghrelin (both at dose of 0.3 mcg/kg bolus i.v.) at 1000 h; (iii) L-arginine (30 gm i.v. over 30 min from 0930 h to 1000 h) followed by GHRH (0.3 μg/kg bolus i.v.) at 1000 h; (iv) L-arginine infusion (30 gm i.v. over 30 min from 0930 h to 1000 h) followed by Ghrelin (0.3 μg/kg bolus i.v.) at 1000 h.
  **Ghrelin dosage is based on 70 kg subject.Total exposure of Ghrelin will be 42 mcg total dose for 2 subject visits (21 mcg per visit).

SUMMARY:
Participants are being asked to take part in this research study to learn why growth hormone(GH) levels decline when estrogen production falls at the time of menopause. GH is a hormone released from the pituitary gland that affects bone, muscle, and fat. Estrogen is a female hormone. Doctors believe that lower estrogen is one of the reasons that GH diminishes in postmenopausal women. However, estrogen does not fall completely. This raises the question whether the little bit of estrogen that is left is doing anything. Lack of GH makes bones thinner, muscles weaker, and fat stores larger. To learn whether the low amount of the body's own estrogen maintains GH secretion after menopause, the investigators need to stop any estrogen you might be taking and then partially block the effect, if any, of your own estrogen. The investigators will use a new estrogen-blocking drug (fulvestrant). Fulvestrant(which also goes by the tradename, Faslodex) was recently approved by the Food and Drug Administration (FDA) to treat breast cancer. Fulvestrant is being used in a non-FDA approved manner in this study (not to treat breast cancer, but to study the effect on Growth Hormone secretion). The drug interferes with how estrogen works in the body, except in the brain. The study that you are considering now tests whether your own estrogen works outside the brain to maintain GH secretion in postmenopausal women. This concept is important, because the brain controls how the pituitary gland secretes GH.

DETAILED DESCRIPTION:
Hypotheses: Endogenous estrogen concentrations contribute significantly to maintaining postmenopausal growth-hormone (GH) secretion and; (b) systemic vis-à-vis CNS actions of endogenous estrogen differentially control the outflow of somatotropic hormones (viz., GH, IGF-I, IGFBP-1).

Approach: contrast regulation of the GH axis in postmenopausal women pretreated with the CNS-excluded selective estrogen-receptor antagonist, fulvestrant, versus placebo.

Background: fulvestrant was released recently by the FDA for therapy of estrogen-sensitive postmenopausal breast cancer. The drug acts as a mechanistically novel inhibitor of estradiol-receptor dimerization, thereby depleting nuclear estrogen receptors. Fulvestrant does not gain access to the CNS. Thus, inhibition of estrogen action will be restricted to non hypothalamic sites of GH-axis control, such as the pituitary gland, liver and fat cells. In contrast, endogenous estrogens have access to both CNS and peripheral sites.

Premise: selective blockade of peripheral estradiol receptors will reduce GH secretion if endogenous estrogens maintain GH secretion via systemic effects.

ELIGIBILITY:
Inclusion Criteria:

* healthy postmenopausal women (ages 50 to 80 y), wherein menopause is defined by the absence of spontaneous menses for 1 y and a serum concentration of FSH > 30 IU/L and of (ultrasensitive) estradiol < 20 pg/mL and verified by medical history and screening blood work;
* normal hemoglobin of >11.0 g/dL in women (a ferritin level will be drawn, and must be normal, if Hgb is 11.0 - 11.5) , Platelets greater than 200 x 109/L, AST 8-48 U/L.
* Subjects (age 50 and above) will have a screening baseline ECG if not on record from the past year.

Exclusion Criteria:

* exposure to psychotropic or neuroactive drug within five biological half- lives;
* undesirability, disinclination or ill advisability of withholding estrogen supplements (e.g. under treatment for symptomatic hot flushes; primary physician recommendation);
* BMI < 19 or > 35
* drug or alcohol abuse; psychosis, depression, mania or anorexia nervosa;
* acute or chronic organ or systemic inflammatory disease;
* endocrinopathy, other than primary thyroidal failure receiving replacement;
* although fulvestrant has no known intrinsic estrogenicity, for safety reasons we include contraindication to short-term estrogen exposure; e.g.,estrogen-sensitive neoplasia, undiagnosed vaginal bleeding, deep-venous thrombosis, stroke or threatened stroke, clinical evidence of atherosclerotic heart disease, including myocardial infarction and/or angina, refractory high blood pressure, severe type IV hyperlipidemia:
* nightshift work or recent transmeridian travel (exceeding 3 time zones within 5 days of admission);
* systemic anticoagulation other than anti platelet therapy (in view of i.m. injections of fulvestrant); history of bleeding diathesis (ie; disseminated coagulation (DIC), clotting factor deficiency
* acute weight change (> 3 kg in 6 weeks); and/or
* unwillingness to provide written informed consent.
* Platelets less than 200 x 109 /L
* International normalization ratio(INR) (Prothrombin time) greater than 1.6
* Total bilirubin greater than 1.5 x ULRR
* ALT or AST greater than 2.5 xULRR if no demonstrable liver metastases or greater
* History or hypersensitivity to active or inactive excipients of fulvestrant (ie; castor oil or Mannitol).

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Veldhuis, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fulvestrant Group: Subjects are given 3 consecutive weekly injections of Fulvestrant 250mg. On days 22-26 after the initial injection, secretagogue combinations are assigned in randomized double-blind order within-subject to include the following conditions:
  (i) L-arginine (30 gm i.v. over 30 min from 0930 h to 1000 h) followed by 5 mL bolus of NS at 1000 h (ii) L-arginine (30 gm i.v. over 30 min from 0930 h to 1000 h) followed by GHRH and Ghrelin (both at dose of 0.3 mcg/kg bolus i.v.) at 1000 h; (iii) L-arginine (30 gm i.v. over 30 min from 0930 h to 1000 h) followed by GHRH (0.3 μg/kg bolus i.v.) at 1000 h; (iv) L-arginine infusion (30 gm i.v. over 30 min from 0930 h to 1000 h) followed by Ghrelin (0.3 μg/kg bolus i.v.) at 1000 h.
- Saline Placebo Group: Subjects are given 3 consecutive weekly injections of saline. On days 22-26 after the initial injection, secretagogue combinations are assigned in randomized double-blind order within-subject to include the following conditions:
  (i) L-arginine (30 gm i.v. over 30 min from 0930 h to 1000 h) followed by 5 mL bolus of NS at 1000 h (ii) L-arginine (30 gm i.v. over 30 min from 0930 h to 1000 h) followed by GHRH and Ghrelin (both at dose of 0.3 mcg/kg bolus i.v.) at 1000 h; (iii) L-arginine (30 gm i.v. over 30 min from 0930 h to 1000 h) followed by GHRH (0.3 μg/kg bolus i.v.) at 1000 h; (iv) L-arginine infusion (30 gm i.v. over 30 min from 0930 h to 1000 h) followed by Ghrelin (0.3 μg/kg bolus i.v.) at 1000 h.
Period: Overall Study
Arm/Group | Fulvestrant Group | Saline Placebo Group
Started | 14 | 16 (1 subject was randomized but withdrew before study interventions.)
Completed | 10 | 14
Not Completed | 4 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects are healthy post-menopausal women from the community.
Groups:
- Saline Group: Subjects are given 3 consecutive weekly injections of Saline. On days 22-26 after the initial injection, secretagogue combinations are assigned in randomized double-blind order within-subject to include the following conditions:
  (i) L-arginine (30 gm i.v. over 30 min from 0930 h to 1000 h) followed by 5 mL bolus of NS at 1000 h (ii) L-arginine (30 gm i.v. over 30 min from 0930 h to 1000 h) followed by GHRH and Ghrelin (both at dose of 0.3 mcg/kg bolus i.v.) at 1000 h; (iii) L-arginine (30 gm i.v. over 30 min from 0930 h to 1000 h) followed by GHRH (0.3 μg/kg bolus i.v.) at 1000 h; (iv) L-arginine infusion (30 gm i.v. over 30 min from 0930 h to 1000 h) followed by Ghrelin (0.3 μg/kg bolus i.v.) at 1000 h.
- Total: Total of all reporting groups
Arm/Group | Fulvestrant Group | Saline Group | Total
Number analyzed (Participants) | 10 | 14 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 9 | 13
  >=65 years | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 14 | 24

OUTCOME MEASURES:

1. Primary Outcome: Mean Baseline GH Concentration
Description: Averaged over 90-min baseline on the saline day.
Time Frame: Withdrawal of blood samples (2.5 mL each) every 10 min for 6 hr. Sampling will begin at 0800 h and conclude at 1400 h.
Measure: Mean (Standard Error); unit: ug/L
Arm/Group | Fulvestrant Group | Saline Placebo Group
Number analyzed (Participants) | 10 | 14
ug/L | 0.23 (0.063) | 0.096 (0.018)
Statistical Analysis 1: Comparison: Fulvestrant Group vs Saline Placebo Group; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Mean GH Concentration (Pulsatile) in Response to Secretagogue
Description: Subjects were administered 4 different secretagogues: (i) L-arginine/Saline, (ii) L-arginine/Ghrelin, (iii) L-arginine/GHRH, and (iv) L-arginine / GHRH + Ghrelin. The result was calculated by averaging values over the 6 hour collection timeframe.
Time Frame: Withdrawal of blood samples (2.5 mL each) every 10 min for 6 hr. Sampling will begin at 0800 h and conclude at 1400 h.
Measure: Mean (Standard Error); unit: ug/L/6h
Arm/Group | Fulvestrant Group | Saline Placebo Group
Number analyzed (Participants) | 10 | 14
ug/L/6h
  Pulsatile GH Response to L-arg/saline | 22.6 (4.1) | 17.3 (3.8)
  Pulsatile GH Response to L-Arg/GHRH | 46.6 (7.1) | 17.4 (7.2)
  Pulsatile GH Response to L-arg/ghrelin | 66.9 (11) | 66.8 (8.8)
  Pulsatile GH Response to L-arg/ghrelin + GHRH | 214 (23) | 178 (27)
Statistical Analysis 1: Comparison: Fulvestrant Group vs Saline Placebo Group; Test type: Superiority or Other; p < 0.05, ANOVA; Two-way ANOVA in a 2x4 factorial nested design with repeated measures

3. Secondary Outcome: Mean Mass of GH Released Per Burst in Response to Secretagogue
Description: Subjects were administered 4 different secretagogues: (i) L-arginine/Saline, (ii) L-arginine/Ghrelin, (iii) L-arginine/GHRH, and (iv) L-arginine / GHRH + Ghrelin. The result was calculated on each 6-hr pool of data by utilizing a previously published deconvolution method and analyzed via two-way ANOVA.
Time Frame: Withdrawal of blood samples (2.5 mL each) every 10 min for 6 hr. Sampling will begin at 0800 h and conclude at 1400 h.
Measure: Mean (Standard Error); unit: ug/L
Arm/Group | Fulvestrant Group | Saline Placebo Group
Number analyzed (Participants) | 10 | 14
ug/L
  Mean Mass of GH per Burst post L-Arg/Saline | 12.6 (2.9) | 7.5 (1.8)
  Mean Mass of GH per Burst post L-Arg/GHRH | 48.4 (7.5) | 44.4 (8.9)
  Mean Mass of GH per Burst post L-Arg/Ghrelin | 64.7 (12) | 45.5 (8.7)
  Mean Mass of GH per Burst post L-Arg/GHRH+Ghrelin | 203 (25) | 164 (29)
Statistical Analysis 1: Comparison: Fulvestrant Group vs Saline Placebo Group; Test type: Superiority or Other; p < 0.05, ANOVA — Unit of "mass secreted per burst" is in ug/L. An automated deconvolution method was used and mathematically verified by direct statistical proof and empirically validated using hypothalamopituitary sampling and a simulated pulsatile time series; Two-way ANOVA in a 2x4 factorial nested design with repeated measures

4. Secondary Outcome: Mean Duration of GH Bursts (Mode) in Response to Secretagogue
Description: as for outcome 3
Time Frame: Withdrawal of blood samples (2.5 mL each) every 10 min for 6 hr. Sampling will begin at 0800 h and conclude at 1400 h.
Measure: Mean (Standard Error); unit: min
Arm/Group | Fulvestrant Group | Saline Placebo Group
Number analyzed (Participants) | 10 | 14
min
  Mean Duration of GH Bursts post L-Arg/Saline | 18.0 (0.91) | 16.3 (1.4)
  Mean Duration of GH Bursts post L-Arg/GHRH | 17.6 (0.45) | 15.4 (0.88)
  Mean Duration of GH Bursts post L-Arg/Ghrelin | 12.8 (1.1) | 12.7 (1.0)
  Mean Duration of GH Bursts post L-Arg/GHRH+Ghrelin | 12.7 (0.92) | 12.8 (0.80)
Statistical Analysis 1: Comparison: Fulvestrant Group vs Saline Placebo Group; Test type: Superiority or Other; p < 0.05, ANOVA; Two-way ANOVA in a 2x4 factorial nested design with repeated measures

5. Secondary Outcome: Mean GH Half-Life in Response to Secretagogue
Description: as for outcome 3
Time Frame: Withdrawal of blood samples (2.5 mL each) every 10 min for 6 hr. Sampling will begin at 0800 h and conclude at 1400 h.
Measure: Mean (Standard Error); unit: min
Arm/Group | Fulvestrant Group | Saline Placebo Group
Number analyzed (Participants) | 10 | 14
min
  Mean GH Half-life duration post L-Arg/Saline | 15.4 (1.1) | 15.0 (0.84)
  Mean GH Half-life duration post L-Arg/GHRH | 17.2 (0.59) | 17.5 (0.70)
  Mean GH Half-life duration post L-Arg/Ghrelin | 19.4 (0.3) | 19.0 (0.35)
  Mean GH Half-life duration post L-Arg/GHRH+Ghrelin | 19.0 (0.53) | 19.1 (0.48)
Statistical Analysis 1: Comparison: Fulvestrant Group vs Saline Placebo Group; Test type: Superiority or Other; p < 0.05, ANOVA; Two-way ANOVA in a 2x4 factorial nested design with repeated measures

ADVERSE EVENTS:
Time Frame: Total adverse event data for the study was collected from 2009-2013 - or the duration of the study. For each individual, adverse event data was collected over approximately one month.
Arm/Group | Fulvestrant Group | Saline Placebo Group
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/15
Other Adverse Events (participants affected / at risk) | 2/14 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant Group (N=14) | Saline Placebo Group (N=15)
Vasovagal reaction with syncope (Surgical and medical procedures) | 1 | 0 — Subject had a syncopal episode while on her way home after a study visit.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant Group (N=14) | Saline Placebo Group (N=15)
Generalized malaise (Surgical and medical procedures) | 1 | 0
Erythema post Fulvestrant injections (Surgical and medical procedures) | 1 | 0 — Developed small 3-4cm erythematoses on bilateral wrists/forearms 3 days after Fulvestrant injection

LIMITATIONS AND CAVEATS:
Strengths and limitations of the study include the potentially confounding effects of body composition (not studied here except at the level of BMI), underlying physical fitness of subjects, size of the cohort, and the brevity of the study (2 months)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes